CLINICAL TRIAL: NCT02419248
Title: Dermatological Evaluation of Topical Compatibility, Primary Skin Irritability, Accumulated Skin Irritability, and Dermal Sensitisation
Acronym: DERM EV TOPIC
Status: Completed | Type: Observational
Sponsor: Kley Hertz S/A (Industry)
Responsible Party: Sponsor
Other Study IDs: KLEY HERTZ-001
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Skin Irritability

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Check the safety under normal conditions of use through the verification of emergence signs of irritability and sensitisation of the genital mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 70 years old;
* Skin types: I (light caucasian), II (caucasian), III (light dark) and IV (dark)
* intact skin where the product will be applied
* Agreement to comply with the test procedures and attend the clinic in the days and ixed times for medical assessments and application and reading of dressings
* Signature of informed consent form

Exclusion Criteria:

* Pregnancy and lactation
* Use of anti-inflammatory and immunosuppressive drugs from 30 days up to three months prior to selection;
* Diseases that cause immune suppression;
* Personal history of atopy;
* History of sensitisation and irritability to topical products;
* Active cutaneous pathologies (local and / or scattered) that may interfere in the study results;
* Use of new drugs and/or cosmetics during the experiment;
* Skin reactivity;
* Previous participation in a study with the same product under test;
* Volunteers who have congenital or acquired known immunodeficiency;
* Relevant medical history or current evidence of alcohol or other drugs abuse;
* Known historical or suspected intolerance to any ingredient of the product under study (product under test or comparator);
* Sponsor's employees involved in the study, or close family member of an employee involved in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with age from 18 to 70 years old, with skin color varying between clear caucasian to dark.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse effects in maximized conditions | 40 days